CLINICAL TRIAL: NCT03613051
Title: Assessment of Movement Skills in Autism Spectrum Disorder
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Dina Tharwat mohamed ali (Other)
Responsible Party: Sponsor-Investigator, Dina Tharwat mohamed ali, Principal Investigator, Assiut University
Organization: Assiut University (Other)
Other Study IDs: movement skills in autism
Record Dates: First submitted 2018-07-19; First posted 2018-08-02 (Actual); Last update posted 2019-02-26 (Actual); Status verified 2018-07

CONDITIONS: Movement Disorders
MeSH Terms: conditions — Movement Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- age band one: age band one ( from 3 to 6 years ) we test manual dexterity by posting coins with prefered hand and non prefered hand test balance by jumping on mats
  Interventions: Behavioral: Movement Assessment Battery for children
- age band two: age band two ( from 7 to 10 years ) test manual dexterity by threading lace
  Interventions: Behavioral: Movement Assessment Battery for children
- age band three: age band three ( from 11 to 18 years ) test manual dexterity by turning pegs test balance by zigzag hopping
  Interventions: Behavioral: Movement Assessment Battery for children

INTERVENTIONS:
Behavioral: Movement Assessment Battery for children — this test measures manual dexterity , balance , aiming and catching

SUMMARY:
this study is to explore the degree of impairement in movement skills in children with autistic spectrum disorders

DETAILED DESCRIPTION:
Motor impairments in neurodevelopmental disorders specifically autism spectrum disorder (ASD) , are prevalent and pervasive . However ,sensori-motor development and self-care activities such as bathing, dressing, eating and toileting, remain little explored in comparison to the other areas of development. Some children with ASD have difficulty mastering self-care skills, which we will call daily living skills .

ELIGIBILITY:
Inclusion Criteria:

* all children with autism from the age of 3 years to 18 years

Exclusion Criteria:

* children less than 3 years , children with neurodegenerative disorders or cerebral palsy

Ages: 3 Years to 18 Years | Sex: All
Age Groups: Child, Adult
Study Population: children from age of 3 years to 18 years with autism not having other brain disease
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2019-04-01 (Estimated); Primary Completion 2019-12-01 (Estimated); Study Completion 2020-04-01 (Estimated)

PRIMARY OUTCOMES:
assessment of motor skills in autism spectrum disorders through Movement Assessmet Battery for Children test ( M-ABC) , using checklists' method . | baseline
  early detection of motor impairement in child with autism and possbillity of prevention .

REFERENCES:
- [Background] Craig F, Lorenzo A, Lucarelli E, Russo L, Fanizza I, Trabacca A. Motor competency and social communication skills in preschool children with autism spectrum disorder. Autism Res. 2018 Jun;11(6):893-902. doi: 10.1002/aur.1939. Epub 2018 Mar 1. PMID 29493892
- [Background] Purpura G, Fulceri F, Puglisi V, Masoni P, Contaldo A. Motor coordination impairment in children with autism spectrum disorder: a pilot study using Movement Assessment Battery for Children-2 Checklist. Minerva Pediatr. 2020 Feb;72(1):22-29. doi: 10.23736/S0026-4946.16.04633-8. Epub 2016 Oct 12. PMID 27733748